CLINICAL TRIAL: NCT01922765
Title: Evaluation of the Efficacy of Concomitant Therapy for Eradication of Helicobacter Pylori
Brief Title: Concomitant Therapy of H. Pylori
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Collaborators: Bucheon St. Mary's Hospital (Other); St Vincent's Hospital (Other)
Responsible Party: Principal Investigator, Jin Il Kim, MD, PhD, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: concomitant
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Gastritis, Gastric Ulcer, and Duodenal Ulcer
Keywords: Helicobacter; Eradication
MeSH Terms: conditions — Gastritis; Stomach Ulcer; Duodenal Ulcer | interventions — Amoxicillin; Clarithromycin; Metronidazole; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- AOC group (Experimental): AOC group: treated with amoxicillin, rabeprazole, clarithromycin for 7 days
  Interventions: Drug: amoxicillin, clarithromycin, metronidazole, rabeprazole
- AOM group (Experimental): AOM group: treated with amoxicillin, rabeprazole, metronidazole for 7 days
  Interventions: Drug: amoxicillin, clarithromycin, metronidazole, rabeprazole
- Sequential group (Experimental): Sequential group: treated with amoxicillin, rabeprazole for 5 day, followed by clarithromycin, metronidazole, rabeprazole for 5 days
  Interventions: Drug: amoxicillin, clarithromycin, metronidazole, rabeprazole
- concomitant group (Experimental): concomitant group: treated with amoxicillin, clarithromycin, metronidazole, rabeprazole for 7 days
  Interventions: Drug: amoxicillin, clarithromycin, metronidazole, rabeprazole

INTERVENTIONS:
Drug: amoxicillin, clarithromycin, metronidazole, rabeprazole
  Other Names: AOC group: treated with amoxicillin, rabeprazole, clarithromycin for 7 days; AOM group: treated with amoxicillin, rabeprazole, metronidazole for 7 days; Sequential group: treated with amoxicillin, rabeprazole for 5 day, followed by clarithromycin, metronidazole, rabeprazole for 5 days; concomitant group: treated with amoxicillin, clarithromycin, metronidazole, rabeprazole for 7 days

SUMMARY:
If we compare eradication rate of Helicobacter pylori divided to 4 groups: amoxicillin, rabeprazole, clarithromycin(AOC), amoxicillin, rabeprazole, metronidazole(AOM), treated with amoxicillin, rabeprazole for 5 day, followed by clarithromycin, metronidazole, rabeprazole for 5 days(sequential), amoxicillin, clarithromycin, metronidazole, rabeprazole(concomitant), then the eradication rate of concomitant group will be the highest.

DETAILED DESCRIPTION:
* Subject: The patient of gastritis, gastric ulcer, and duodenal ulcer infected with Helicobacter pylori
* 170 subjects per group
* Eradication regimens are as follows: AOC group, treated with amoxicillin, rabeprazole, clarithromycin for 7 days; AOM group, treated with amoxicillin, rabeprazole, metronidazole for 7 days; sequential group, treated with amoxicillin, rabeprazole for 5 day, followed by clarithromycin, metronidazole, rabeprazole for 5 days; concomitant group, treated with amoxicillin, clarithromycin, metronidazole, rabeprazole for 7 days

ELIGIBILITY:
Inclusion Criteria:

* patients infected with Helicobacter pylori

Exclusion Criteria:

* cancer
* pregnancy
* formerly treated with eradication

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of concomitant therapy for eradication of Helicobacter pylori | 6 months (Feb 2014)
  measure eradication rate of H.pylori with urea breath test(UBT) after 6 to 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Yeouido St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee HJ, Kim JI, Lee JS, Jun EJ, Oh JH, Cheung DY, Chung WC, Kim BW, Kim SS. Concomitant therapy achieved the best eradication rate for Helicobacter pylori among various treatment strategies. World J Gastroenterol. 2015 Jan 7;21(1):351-9. doi: 10.3748/wjg.v21.i1.351. PMID 25574111